CLINICAL TRIAL: NCT01913171
Title: Effect of Hula Hooping as Compared to Walking on Adipose Tissue Distribution, Metabolic Parameters and Adipose Tissue Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Sanja Sadevirta, MD, University of Helsinki
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: HULA 233401; HULA233401 (Other: HUS Tietu)
Record Dates: First submitted 2013-06-18; First posted 2013-07-31 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Android Obesity, Metabolic Parameters and Adipose Tissue (AT) Gene Expression
MeSH Terms: conditions — Obesity, Abdominal | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking (Active Comparator): WALK. The participants were instructed to walk daily, at first week 12minutes/day, week II 16mins/day, week III 20mins/day, week IV 24 mins/day, week V 28mins/day, week VI 32mins/day at a pace that would moderately increase heart rate and result in sweating
  Interventions: Other: Exercise
- Hula-hooping (Active Comparator): HULA. The participants were instructed to hula hoop daily, at first week 6minutes/day, week II 8mins/day, week III 10mins/day, week IV 12 mins/day, week V 14mins/day, week VI 16mins/day
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise

SUMMARY:
o determine effects of hula-hooping on android obesity, metabolic parameters and adipose tissue (AT) gene expression.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 70 years
* central adiposity as measured by the waist circumference (>80 cm in females and >94 cm in males) (9)
* ability to hula-hoop for a minimum of 2 minutes and to have the necessary space available for this activity either at home or at work
* ability to communicate meaningfully with the investigator and legal competence to provide written informed consent

Exclusion Criteria:

* clinical or biochemical evidence of disease other than obesity as judged by history, physical examination and standard laboratory tests
* excessive use of alcohol, i.e., over 20 g/day
* use of medications known to affect glucose or lipid metabolism and
* pregnancy or lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Android obesity | 6weeks
  The primary objective was to evaluate the change in the % fat in the android region as measured by DEXA during 6 weeks of HULA as compared to WALK

SECONDARY OUTCOMES:
metabolic parameters | 6weeks
  The secondary objectives included the comparison of differences in waist circumference (cm), relative and absolute trunk and limb muscle mass as measured by DEXA (% and kg), fasting plasma glucose (mmol/l), fasting serum insulin (mU/l), liver enzymes (U/l), fasting plasma LDL and HDL cholesterol and triglycerides (mmol/l). Gene expression was analyzed in adipose tissue biopsies collected before and after each exercise intervention.

OTHER OUTCOMES:
adipose tissue inflammation | 6weeks
  To determine the effects of HULA compared to WALK on adipose tissue inflammation, a needle aspiration biopsy of abdominal s.c. adipose tissue was taken under local anesthesia with lidocaine before and after each exercise intervention. The adipose tissue sample was immediately frozen in liquid nitrogen and then stored at -80°C until analysis. Total RNA from s.c. AT was isolated.Relative quantification for the genes of interest (see list below) was carried out using normalization to the 36B4 and β-actin mRNA values.
  ABCA1 Adiponectin ANGPTL8 CHOP CD4 CD8 CD68 ETFDH FOXP3 GLUT4 MCP-1 MRC-1 PGC-1α VEGF-A β-actin

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Lahelma M, Sadevirta S, Lallukka-Bruck S, Sevastianova K, Mustelin L, Gylling H, Rockette-Wagner B, Kriska AM, Yki-Jarvinen H. Effects of Weighted Hula-Hooping Compared to Walking on Abdominal Fat, Trunk Muscularity, and Metabolic Parameters in Overweight Subjects: A Randomized Controlled Study. Obes Facts. 2019;12(4):385-396. doi: 10.1159/000500572. Epub 2019 Jun 19. PMID 31216547